CLINICAL TRIAL: NCT04251403
Title: A Novel Approach to the Surveillance of Pre-Malignant Gastric Lesions
Brief Title: Novel Approach to Surveillance of Gastric Lesions
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, Monika Laszkowska, Principal Investigator, New York Presbyterian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB-AAAS8330
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Intestinal Metaplasia of Gastric Mucosa; Gastric Dysplasia; Gastric Cancer; Atrophic Gastritis
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic

STUDY DESIGN:
Intervention Model Description: This is a pilot feasibility study. High-risk individuals with known history of gastric precursor lesions (atrophic gastritis, intestinal metaplasia, dysplasia) who are presenting for routine surveillance endoscopy will undergo mucosal irrigation and collection of gastric aspirate for analysis, in addition to standard of care (visual inspection on endoscopy).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mucosal Irrigation (Experimental): Following routine endoscopic evaluation, investigators will utilize the ERBEJET 2 device (ERBE USA Inc), which is commercially available for the treatment of mucosal lesions, to sample cells from the mucosal surface of the stomach. The aspirate will be collected for cytologic/pathologic assessment.
  Interventions: Diagnostic Test: Mucosal Irrigation

INTERVENTIONS:
Diagnostic Test: Mucosal Irrigation — Following routine endoscopic evaluation, investigators will utilize the ERBEJET 2 device (ERBE USA Inc), which is commercially available for the treatment of mucosal lesions, to sample cells from the mucosal surface of the stomach. The aspirate will be collected for cytologic/pathologic assessment.

SUMMARY:
This will be a pilot study investigating the feasibility of using pressurized irrigation of the stomach mucosa to obtain gastric aspirate cell samples for analysis and identification of premalignant lesions of the stomach.

DETAILED DESCRIPTION:
Gastric cancer is an important public health concern, accounting for 26,240 new cases in the United States (US) annually. Outcomes are poor, with 5-year survival of 31%, but improve when lesions are detected at early stages amenable to curative therapy. Research has shown that lesions such as atrophic gastritis and gastric intestinal metaplasia are precursors to more advanced lesions such as dysplasia and adenocarcinoma, thus providing a potential target for early intervention. Gastric cancer screening programs have decreased mortality in high-prevalence countries like Japan. However, providers in low-prevalence settings are less experienced at detecting precursor lesions endoscopically on visual inspection. This pilot study will investigate a novel approach to screening for precursor lesions and early detection of gastric cancer by utilizing pressurized irrigation of the gastric mucosa. The study will target patients with a known history of gastric precursor lesions (atrophic gastritis, intestinal metaplasia, history of dysplasia) who are presenting for routine surveillance endoscopy. Following routine endoscopic evaluation, the investigators will utilize the ERBEJET 2 device (ERBE USA Inc), which is commercially available for the treatment of mucosal lesions, to sample cells from the mucosal surface of the stomach. The aspirate will be collected for cytologic/pathologic assessment. The goal is that this technique will simplify testing for precursor lesions of gastric cancer, making screening more effective in regions of lower prevalence where providers are less experienced with visual identification of such lesions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a known history of gastric precursor lesions (atrophic gastritis, intestinal metaplasia, history of dysplasia) who are presenting for routine surveillance endoscopy

Exclusion Criteria:

* Personal history of gastric cancer
* Personal history of irritable bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Correlation of pathologic diagnosis from gastric aspirate compared with diagnosis from standard endoscopic inspection and biopsies. | Intra-procedural
  Investigators will compare how the diagnosis determined from pathologic/cytologic analysis gastric aspirate samples will compare with diagnosis obtained from standard endoscopic inspection and biopsies. The diagnoses of interest will be normal mucosa, atrophic gastritis, intestinal metaplasia, dysplasia, or malignancy. This will be reported as the percentage of concordant diagnoses.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Lightdale, MD, Principal Investigator — New York Presbyterian - Columbia University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamashima C. Current issues and future perspectives of gastric cancer screening. World J Gastroenterol. 2014 Oct 14;20(38):13767-74. doi: 10.3748/wjg.v20.i38.13767. PMID 25320514
- [Background] Gupta S, Li D, El Serag HB, Davitkov P, Altayar O, Sultan S, Falck-Ytter Y, Mustafa RA. AGA Clinical Practice Guidelines on Management of Gastric Intestinal Metaplasia. Gastroenterology. 2020 Feb;158(3):693-702. doi: 10.1053/j.gastro.2019.12.003. Epub 2019 Dec 6. No abstract available. PMID 31816298
- [Background] Kim GH, Liang PS, Bang SJ, Hwang JH. Screening and surveillance for gastric cancer in the United States: Is it needed? Gastrointest Endosc. 2016 Jul;84(1):18-28. doi: 10.1016/j.gie.2016.02.028. Epub 2016 Mar 3. PMID 26940296
- [Background] BASTOS AL, MADEIRA F. A SIMPLE DEVICE FOR EXFOLIATIVE CYTOLOGY OF THE STOMACH. Gut. 1964 Apr;5(2):192-3. doi: 10.1136/gut.5.2.192. No abstract available. PMID 14159412